CLINICAL TRIAL: NCT01145976
Title: Randomized Comparison of Cyclophosphamide Versus Fludarabine in Addition to Anti-thymocyte Globulin for the Conditioning Therapy in Allogeneic Hematopoietic Cell Transplantation for Adult Acquired Aplastic Anemia
Brief Title: Comparison of Cy-Atg vs Flu-Atg for the Conditioning Therapy in Allo-HCT for Adult Aplastic Anemia
Acronym: CyATG-FluATG
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cooperative Study Group A for Hematology (Network)
Responsible Party: Principal Investigator, Yae Eun Jang, Research nurse, Cooperative Study Group A for Hematology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-021
Record Dates: First submitted 2010-05-19; First posted 2010-06-17 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Aplastic Anemia
Keywords: aplastic anemia, fludarabine, cyclophosphamide, thymoglobulin
MeSH Terms: conditions — Anemia, Aplastic | interventions — Cyclophosphamide; thymoglobulin; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CY-ATG(Arm1) (Active Comparator): Hydration with 0.45% NaCl at 6 liters/24 hours will be started on day -5. Cy 50 mg/kg in D5W 200 ml i.v. over 1-2 hours on days -5 to -2 by pump through a central venous catheter.
  Thymoglobuline 3 mg/kg in N/S 500-800 mL (less than 0.5 mg/mL) or lymphoglobuline 15 mg/kg in N/S 500-800 mL (less than 2 mg/mL) iv daily at 8 am on days -4 to -2
  Interventions: Drug: Cy-ATG
- Flu-ATG(Arm2) (Experimental): Fludarabine 30 mg/m2 will be infused intravenously over 30 minutes in D5W 100 ml for 6 consecutive days (days -7 to -2) Thymoglobuline 3 mg/kg in N/S 500-800 mL (less than 0.5 mg/mL) or lymphoglobuline 15 mg/kg in N/S 500-800 mL (less than 2 mg/mL) iv daily at 8 am on days -4 to -2
  Interventions: Drug: Flu-ATG

INTERVENTIONS:
Drug: Cy-ATG — Hydration with 0.45% NaCl at 6 liters/24 hours will be started on day -5. Cy 50 mg/kg in D5W 200 ml i.v. over 1-2 hours on days -5 to -2 by pump through a central venous catheter.
  Thymoglobuline 3 mg/kg in N/S 500-800 mL (less than 0.5 mg/mL) or lymphoglobuline 15 mg/kg in N/S 500-800 mL (less than 2 mg/mL) iv daily at 8 am on days -4 to -2
  Other Names: Cyclophosphamide; Thymoglobulin
  Arms: CY-ATG(Arm1)
Drug: Flu-ATG — Fludarabine 30 mg/m2 will be infused intravenously over 30 minutes in D5W 100 ml for 6 consecutive days (days -7 to -2) Thymoglobuline 3 mg/kg in N/S 500-800 mL (less than 0.5 mg/mL) or lymphoglobuline 15 mg/kg in N/S 500-800 mL (less than 2 mg/mL) iv daily at 8 am on days -4 to -2
  Other Names: Fludarabine; Thymoglobulin
  Arms: Flu-ATG(Arm2)

SUMMARY:
The purpose of this study is to reduce the regimen related toxicities and transplantation related mortality after allogeneic stem cell transplantation in adult acquired aplastic anemia (AA), the trials of reduced dose of Cy along with fludarabine and ATG were performed.11-21 The investigators preliminary data of randomized comparison of cyclophosphamide plus fludarabine versus cyclophosphamide alone in addition to anti-thymocyte globulin for the conditioning therapy in allogeneic hematopoietic cell transplantation for bone marrow failure syndrome supports reduced dose of Cy along with fludarabine and ATG.

Conditioning regimen without Cy may reduce RRT because Cy-containing conditioning remains several RRT such as hemorrhagic cystitis, SOS and graft versus host disease (GvHD). Recently there were small trials of fludarabine and ATG (Flu-ATG) for the conditioning regimen of alloHSCT.22-24 These data raised the feasibility of fludarabine and ATG without Cy for patients with AA.

This new conditioning regimen of Flu-ATG will be compared to standard regimen of Cy- ATG in a randomized controlled trial.

DETAILED DESCRIPTION:
TREATMENT PLAN

* The patients will be admitted to laminar air flow room.
* The patients will have triple lumen Hickman central venous catheter (CVC) placed. Chest X-ray should be taken after CVC placement to confirm the location of CVC and absence of pneumothorax.
* Menstruating women will be given norethindrone (Primolut) 10 mg po daily.

  1. The preparatory regimen is as follows:

     Conditioning therapy will start on day -5 in patients who are randomized to receive Cy+ATG. Hydration with 0.45% NaCl at 6 liters/24 hours will be started on day -5. Cy 50 mg/kg in D5W 200 ml i.v. over 1-2 hours on days -5 to -2 by pump through a central venous catheter. Mesna 12 mg/kg iv push immediately before Cy and 3, 6, 9, and 12 hours after Cy. Thymoglobuline 3 mg/kg in N/S 500-800 mL (less than 0.5 mg/mL) or lymphoglobuline 15 mg/kg in N/S 500-800 mL (less than 2 mg/mL) iv daily at 8 am on days -4 to -2. Premedication for ATG (ALG) will include methylprednisolone 2 mg/kg iv infusion, Tylenol 600 mg po, and Avil 45.5 mg iv push. The doses of cyclophosphamide and ATG (ALG) will be calculated using actual body weight.

     Conditioning therapy will start on day -7 in patients who are randomized to receive Flu-ATG. Fludarabine 30 mg/m2 will be infused intravenously over 30 minutes in D5W 100 ml for 6 consecutive days (days -7 to -2). Thymoglobuline 3 mg/kg in N/S 500-800 mL (less than 0.5 mg/mL) or lymphoglobuline 15 mg/kg in N/S 500-800 mL (less than 2 mg/mL) iv daily at 8 am on days -4 to -2. Premedication for ATG (ALG) will include methylprednisolone 2 mg/kg iv infusion, Tylenol 600 mg po, and Avil 45.5 mg iv push. The doses of cyclophosphamide and ATG (ALG) will be calculated using actual body weight.
  2. GVHD prophylaxis will include cyclosporine plus methotrexate.

     The patients will receive cyclosporine 1.5 mg/kg in NS 100 ml i.v. over 2-4 hours q 12 hrs (dose of cyclosporine rounded to nearest 5 mg) starting day -1 at 6 a.m. Cyclosporine dose will be adjusted to provide appropriate level and according to the change of renal function (see Appendix II).

     Cyclosporine dosing will be changed to oral dosing when oral feeding became feasible at the twice the i.v. dosages.

     In addition, the patients will receive methotrexate 15 mg/m2 i.v. push on day 1 and 10 mg/m2 on days 3, 6, and 11. The dose of methotrexate will be decreased or omitted according to the guideline provided in Appendix III.

     The dose of cyclosporine will be decreased by 10 % every month starting day 60 of BMT provided that there is no clinical evidence of GVHD.
  3. Hematopoietic stem cell collection from the donors.

Mobilized peripheral blood stem cells are used but bone marrow collection in case of sibling donor is permitted.

Bone marrow collection

* Packed red cell 2 units will be collected from donor for autologous transfusion before hematopoietic stem cells collection.
* Hematopoietic stem cells are collected from bone marrow under an appropriate anesthesia.
* After collection, Feroba 1T bid will be given to the donor for 1 month.

Mobilized peripheral blood stem cell collection

* Recombinant human granulocyte colony-stimulating factor (G-CSF) 10 mcg/kg will be administered sc to stem cell donors daily for 4 days (from day -3 to day 0).
* Daily CBC will be done.
* Starting day 4 of G-CSF administration (day 0), peripheral blood mononuclear cells will be collected by leukapheresis CS3000 for 2 days (days 0 and 1). A sample will be taken for cell count of total cell, mononuclear cells, CD34+ cell, CD3+ cell, CD4+ cells, and CD8+ cells.
* After the sampling, the final product will be infused to the patients immediately on day 0 and day1.
* At least 2x10^6/kg of CD34+ cells should be collected on day 0. If not, additional collection may be scheduled under the discretion of attending physician.

  4.Hematopoietic stem cell infusion
* For ABO matched or minor mismatched transplantation, premedication with Avil 45.5 mg i.v. push and tylenol 600 mg p.o. will be given. Stem cell will be infused via CVC over 1 hr.
* For major ABO mismatched transplantation, premedication with Avil 45.5 mg i.v. push, tylenol 600 mg p.o., 10 % mannitol 100 g i.v. over 4 hrs will be started 30 min before stem cell infusion, and hydrocortisone 250 mg i.v. will be given immediately before and 30 min of stem cell infusion. Stem cells will be infused via CVC over 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Severe aplastic anemia
* Severe aplastic anemia (SAA) is defined as a hypocellular bone marrow (cellularity<25%) and two or more of the following: granulocyte count <500/ml, platelet count <20,000/ml, and corrected reticulocyte count <1.0%
* Very severe aplastic anemia (VSAA) is defined as the criteria for SAA plus a granulocyte count <200/ml
* Patients should be 15 years of age or older, but younger than 65 years.
* The performance status of the patients should be 70 or over by Karnofsky performance scale (see Appendix I).
* Patients must have adequate hepatic function (bilirubin less than 2 mg/dl, AST and ALT less than three times the upper normal limit)
* Patients must have adequate renal function (creatinine less than 2.0 mg/dl).
* Patients must have adequate cardiac function (ejection fraction > 45% on echocardiogram).

Exclusion criteria:

* Patients should not have major illness or organ failure.
* Patients must not have a psychiatric disorder or mental deficiency severe as to make compliance with the treatment unlikely, and making informed consent impossible.
* Patients must not be in pregnancy.
* Hypoplastic myelodysplastic syndrome
* Paroxysmal nocturnal hemoglobinuria

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2010-03; Primary Completion 2015-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
regimen-related toxicities(RRT) | 7 years
  * The RRTs will be evaluated in terms of mucositis, hemorrhagic cystitis, SOS, acute graft versus host disease (GvHD), infection rate, graft failure, time to engraftment.
  * Overall feasibility will be evaluated by RRTs, time to engraftment, chronic GvHD, treatment-related mortality (TRM), relapse rate, infertility, chimerism status, changes of hemostatic variables, event-free survival and overall survival.

SECONDARY OUTCOMES:
Overall feasibility | 7 years
  Day 100 mortality rate, overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Hawk Kim, professor, Principal Investigator — Ulsan University Hospital, University of Ulsan College of Medicine
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

REFERENCES:
- [Derived] Kim H, Lee JH, Joo YD, Bae SH, Hyun MS, Lee JH, Kim DY, Lee WS, Ryoo HM, Kim MK, Park JH, Lee KH; Cooperative Study Group A for Hematology (COSAH). A randomized comparison of cyclophosphamide vs. reduced dose cyclophosphamide plus fludarabine for allogeneic hematopoietic cell transplantation in patients with aplastic anemia and hypoplastic myelodysplastic syndrome. Ann Hematol. 2012 Sep;91(9):1459-69. doi: 10.1007/s00277-012-1462-x. Epub 2012 Apr 18. PMID 22526363
- See also: Randomized comparison of cyclophosphamide versus fludarabine in addition to anti-thymocyte globulin for the conditioning therapy in allogeneic hematopoietic cell transplantation for bone marrow failure syndrome — http://www.google.co.kr